CLINICAL TRIAL: NCT05398601
Title: Effects Of Periosteal Electrical Dry Needling In Patients With Knee Osteoarthritis
Brief Title: Periosteal Electrical Dry Needling in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01209 Mudassar
Record Dates: First submitted 2022-04-21; First posted 2022-06-01 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
Keywords: Dry needling; Acupuncture; Mobilization with movement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Movement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOBILIZATION WITH MOVEMENT (Active Comparator): MOBILIZATION with MOVEMENT
  TENS, MWM techniques for Knee
  Interventions: Other: MOBILIZATION with MOVEMENT
- periosteal electrical dry needling (Experimental): TENS, periosteal electrical dry needling 4 point technique for Knee
  Interventions: Other: Periosteal electrical dry needling

INTERVENTIONS:
Other: MOBILIZATION with MOVEMENT — They would be receiving conventional treatment as follow:
  TENS (Transcutaneous electrical nerve stimulation) applied asymmetrical, biphasic waveform, pulse duration at 100 ms, intensity 10 percent below the motor threshold - 10 mins Hot Pack - 10 mins ULTRASOUND - 10 mins
  Additionally, the would receive MWM techniques for Knee
  1. Medial glide
  2. Medial+ Internal rotation glide
  3. Lateral Glide+ Internal Rotation glide
  4. Anterior glide
  5. Posterior glide
  Arms: MOBILIZATION WITH MOVEMENT
Other: Periosteal electrical dry needling — They would be receiving conventional treatment as follow:
  TENS (asymmetrical, biphasic waveform, pulse duration at 100 ms, intensity 10 percent below the motor threshold) - 10 mins HOT PACK - 10 mins ULTRASOUND - 10 mins
  Additionally, the would receive periosteal electrical dry needling 4 point technique for Knee
  Four sterile, single-use 30-gauge dry needles would be inserted into the following locations of the symptomatic knee(s) until they touch bone:
  1. Medial femoral condyle
  2. Lateral femoral condyle
  3. Flare of the tibia
  4. Head of the fibula Needles would be stimulated with 100 Hz for 30 minutes. The intensity of the stimulus would be adjusted so that it would be clearly felt but would not cause discomfort. The stimulus intensity would be adjusted periodically so that it is perceptible for the entire 30 minutes of PST.
  Arms: periosteal electrical dry needling

SUMMARY:
To determine the effect of periosteal electrical dry needling as an adjuvant to MWM in knee osteoarthritis for pain management, for improvement in functional activities and for ROM (Range Of Motion)

DETAILED DESCRIPTION:
Periosteal stimulation therapy (PST) or periosteal electroacupuncture applies direct electrical stimulation of the periosteum and its associated nerves using parsimoniously applied acupuncture needles over bony prominences. It is an aggressive local treatment for deep pain problems such as OA (osteoarthritis ) .

Mobilization with movement (MWM) is a manual therapy technique that is used most frequently for the management of musculoskeletal conditions. In this technique, the physiological movement is performed in a pain-free manner with accessory glides being applied in the direction towards the opposite of the previously painful movement to have the greatest improvement MWMs has shown promising various therapeutic benefits such as reduction of pain and improved range of motion. Previous evidence has shown the effectiveness of MWM on pain reduction and functional improvement in patients with knee OA.

The rationale for the use of PST in comparison with MWM techniques is to determine the effectiveness of periosteal electrical dry needling for the common use intervention for knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Age group >40,
2. Patient who met American college of Rheumatology criteria of Osteoarthritis,
3. Chronic knee pain > 3 months,
4. Morning stiffness <30 mins,
5. Crepitation
6. Bony tenderness

Exclusion Criteria:

1. Diagnosed Meniscal injury or Ligamentous injury,
2. History of Intraarticular injection in last 3 months,
3. generalized low back related leg pain,
4. Patients with fear of needles,
5. Patients administered with corticosteroids or receiving any other invasive treatment such as PRP, Stem cell therapy, Ozone therapy
6. History of any surgery of lower extremity in last 6 months
7. Malignancy

Ages: 41 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-07-08 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
WOMAC scale for osteoarthritis | 4 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  * Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright
  * Stiffness (2 items): after first waking and later in the day
  * Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties
  The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  Scores range from 0 to 96 for the total WOMAC where 0 represents the best health status and 96 the worst possible status. The higher the score, the poorer the function.

SECONDARY OUTCOMES:
NPRS | 4 weeks
  The NPRS is a segmented numeric version of the visual analog scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
  The scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
6 min walk test | 4 weeks
  The Six-minute walk (6MW) is short walk tests commonly used to evaluate functional recovery after total knee arthroplasty (TKA).
  The object of the test is to walk as far as possible for six minutes. You will walk at your normal pace to a chair or cone, and turn around. And you continue to walk back and forth for six minutes. Time measurement will determine the functional recovery.
Stair climb test | 4 week
  The stair climb test (also known as stair climb power test) is a clinically relevant, safe, and inexpensive field-based assessment of lower body strength, power, and physical function for older adults Stairs (8 - 14 steps) with handrails, stopwatch. Where possible, the 9-step stair test with 20cm (8 inch) step height (range 16-20 cm) and handrail is recommended. 2 mins are required to complete and score,
Range of Motion | 4 week
  A goniometer is an instrument that measures the available range of motion at a joint.
  Normal range of motion, using the anatomical position as zero degrees. Flexion = 0 to 140 degrees. Extension - zero degrees = full extension.

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — RIPHAH INTERNATIONAL UNIVERSITY,ISLAMABAD,PAKISTAN
Locations (1):
- Athlean Physical Therapy Clinic, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No